CLINICAL TRIAL: NCT02071901
Title: A Single Arm, Phase II Study of Eltrombopag to Enhance Platelet Count Recovery in Elderly Patients With Acute Myeloid Leukemia Undergoing Remission Induction Therapy
Brief Title: Eltrombopag Olamine in Improving Platelet Recovery in Older Patients With Acute Myeloid Leukemia Undergoing Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4913; NCI-2014-00252 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (eltrombopag olamine) (Experimental): Patients receive eltrombopag olamine by mouth (PO) daily (QD) until platelet counts reach >= 50,000/uL or for 8 weeks, whichever comes earlier. Treatment continues in the absence of unacceptable toxicity.
  Interventions: Drug: eltrombopag olamine

INTERVENTIONS:
Drug: eltrombopag olamine — Given PO
  Other Names: Promacta; SB 497115; SB-497115; SB497115

SUMMARY:
This phase II trial studies how well eltrombopag olamine works in improving the recovery of platelet counts in older patients with Acute Myeloid Leukemia (AML) undergoing induction (the first treatment given for a disease) chemotherapy. Platelet counts recover more slowly in older patients, leading to risk of complications and the delay of post-remission therapy. Eltrombopag olamine may cause the body to make platelets after chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I.To determine whether eltrombopag leads to early platelet recovery in older AML patients (≥ 60years) who attain morphologic remission on day 14 (range, day 14-17) bone marrow assessment following remission induction chemotherapy (IC).

SECONDARY OBJECTIVES:

I. To determine the effect of eltrombopag on megakaryopoiesis - median time to reach platelet count ≥50,000 /μL and ≥100,000 /μL, number of days of platelet transfusion, rates of platelet transfusion-independence and the median time to reach platelet transfusion independence.

II. To determine the effect of eltrombopag on the rates of clinically significant bleeding events (CSBE).

III. To determine the effect of eltrombopag on erythropoiesis the median time to red blood cell transfusion independence.

IV. To determine the effect of eltrombopag on granulopoiesis- the time taken to reach an absolute neutrophil count of ≥ 500 /μL. V. To determine the safety and tolerability of eltrombopag in AML patients undergoing remission IC - incidence and severity of eltrombopag-related adverse events. VI. To determine rates of complete remission (CR), rates of partial complete remission (CRp), time to attain CR, and time to initiation of post-remission consolidation therapy.

OUTLINE:

Participants receive eltrombopag olamine orally (PO) once daily (QD) until platelet counts reach ≥50,000/uL or for 8 weeks, whichever comes earlier. Treatment continues in the absence of unacceptable toxicity.

After completion of study treatment, participants are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* All categories of AML will be included except for acute promyelocytic leukemia (APL), acute megakaryocytic leukemia, and acute leukemias of ambiguous lineage undergoing 7 + 3 remission IC with cytarabine and an anthracycline (daunorubicin or idarubicin). All cases have to be histopathologically confirmed by a diagnostic bone marrow biopsy. Use of granulocyte colony-stimulating factor (G-CSF) for any indication must have been discontinued at least 7 days prior to entry into the study.
* Patients with secondary AML arising out of Myelodysplastic syndrome (MDS) (all subtypes under WHO [World Health Organization] classification), chronic myelomonocytic leukemia (CMML); therapy-related AML and those with a prior autologous hematopoietic cell transplantation are eligible.
* No morphological evidence of disease on day 14 bone marrow examination following IC
* Must be able to give voluntary informed written consent to participate in the study; informed consent will be obtained prior to initiation of remission IC and before any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment. All men and women of childbearing potential must use acceptable methods of birth control throughout the study as described below:

  1. Females of childbearing potential: Recommendation is for 2 effective contraceptive methods during the study. Adequate forms of contraception are double-barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation.
  2. Male patients with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, during the study or to abstain.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that, in the view of the treating physician, would place the participant at an unacceptable risk if he or she were to participate in the study or would prevent that person from giving informed consent
* Any active malignancy (unrelated, non-hematological malignancy) diagnosed within the past 12 months of starting the study drug (other than curatively treated carcinoma-in-situ of the cervix or non-melanoma skin cancer).
* Secondary AML arising out of myeloproliferative neoplasms [as per the revised 2008 WHO classification of myeloid neoplasms and acute leukemias] and MDS/myeloproliferative disease (MPD) neoplasms other than CMML [as per the revised 2008 WHO classification of myeloid neoplasms and acute leukemias]. Refractory Anemia with Ringed Sideroblasts with thrombocytosis (RARS-T) classified as MDS/MPN neoplasm, unclassifiable will be excluded. AML patients with presenting features suspicious of underlying unrecognized MPD such as marked splenomegaly (> 20 cm) and thrombocytosis (>400,000 per microliter) will be excluded. Patients with relapsed or refractory AML will be excluded.
* Radiation therapy, cytotoxic chemotherapy, and combined modality (both radiation and chemotherapy) used to treat other cancers or medical conditions and administered within 12 months prior to signing informed consent. Use of hydroxyurea or emergent leukapheresis (for cytoreduction of highly elevated white blood cell counts) is permissible. Those AML patients who initially receive treatment with all-trans retinoic acid (ATRA) for presumptive diagnosis of APL but if APL is ruled out in final pathology will be eligible for the study.
* Prior history of treatment with recombinant thrombopoietin (TPO) or TPO-receptor (R) agonists
* History of arterial or venous thrombosis [excluding line-thrombosis] within the last 1 year, or those with known inherited coagulopathies. Arterial or venous thrombosis includes pulmonary embolism, deep vein thrombosis of both upper [excluding line-thrombosis] and lower extremities, coronary artery disease managed medically or requiring intervention (percutaneous stent placement or coronary bypass surgery), cerebrovascular accident (for transient ischemic attacks clinical documentation is required), or involvement of other organs (such as hepatic, renal, spleen or other sites).
* Evidence of fibrosis on bone marrow examination at the time of diagnosis
* Active participation in any other investigational treatment study
* Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure, cardiac arrhythmia, unstable angina or renal insufficiency (acute or chronic) on hemodialysis
* Liver enzymes (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) can not be greater than or equal to 2.5 times the upper limits of normal (ULN)
* Total bilirubin ≥ 1.5 x ULN within 14 days of enrollment.
* Serum creatinine should be ≥ 2.5 x ULN within 14 days of enrollment
* A known immediate or delayed hypersensitivity reaction or idiosyncrasy that, in the opinion of the Medical Monitor is due to drugs chemically related to eltrombopag or excipients (e.g. mannitol)
* Known history of human immunodeficiency virus (HIV) or active hepatitis B or C
* No major surgery within 2 weeks prior to trial enrollment
* Female subject is pregnant or breast-feeding
* Male and female patients who are fertile who do not agree to use an effective barrier methods of birth control (i.e. abstinence) to avoid pregnancy while receiving study treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2023-09-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sudipto Mukherjee, MD, PhD, MPH, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Supportive Care (Eltrombopag Olamine): Patients receive eltrombopag olamine PO QD until platelet counts reach >= 50,000/uL or for 8 weeks, whichever comes earlier. Treatment continues in the absence of unacceptable toxicity.
  eltrombopag olamine: Given PO
Period: Overall Study
Arm/Group | Supportive Care (Eltrombopag Olamine)
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who went on study
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: Years] | 67 [60 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Median Platelet Count >= 50,000/uL
Description: Number of participants with a median platelet count >= 50,000/uL
Time Frame: Day 24 of Treatment
Population: Participants who completed study
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
Participants | 30

2. Secondary Outcome: Median Time Needed to Reach Platelet Count >= 50,000 /µL in Days
Description: Defined as the average number of days from the first day of eltrombopag until the first of five consecutive days with platelet counts >= 50,000 /µL without a platelet transfusion. The time will be summarized using the Kaplan-Meier method and will use the logrank test and proportional hazards models.
Time Frame: up to 12 weeks
Population: Participants who completed study. Statistical tests were not completed because a) Difficulty in obtaining accurate information on the reasons for platelet transfusion in the historical cohort and b) Several participants had platelet counts higher than threshold for starting transfusion, making comparisons not meaningful
Measure: Median (Full Range); unit: days
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
days | 7 [6 to 8]

3. Secondary Outcome: Median Days of Platelet Transfusions
Description: Defined as the median number of days from the first day of eltrombopag until the patient stopped treatment. The time will be summarized using the Kaplan-Meier method and will use the log-rank test and proportional hazards models.
Time Frame: Up to 12 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
days | 10 [8 to 11]

4. Secondary Outcome: Rates of Clinically Significant Bleeding Events
Description: The number of bleeding events experienced by patients during treatment including hematuria, gastrointestinal bleed (with or without requiring intervention, retroperitoneal bleeding, intra-cranial bleed, epistaxis not controlled by conservative measures and muscle or soft tissue hematomas.
Time Frame: Up to 12 weeks
Population: Participants who completed study
Measure: Number; unit: events
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
events | 0

5. Secondary Outcome: Median Time to Absolute Neutrophil Recovery, Defined as > 500/uL
Description: The average number of days patients take to reach a neutrophil count >500/ul as summarized using the Kaplan-Meier method and modeled using logrank test and proportional hazards.
Time Frame: Up to 12 weeks
Population: Data not collected - daily blood counts were not checked once participants were discharged or received post-remission therapy and subsequent follow ups locally
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 0

6. Secondary Outcome: Median Rise in Hemoglobin Level in Patients With Pretreatment Hemoglobin of < 8 g/dL
Description: The median increase in hemoglobin levels in g/dL among patients with a starting hemoglobin level <8g/dL
Time Frame: Up to 12 weeks
Population: as for outcome 5
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 0

7. Secondary Outcome: Complete Response Rate
Description: The percent of participants with a sustained improvement of platelet counts (independent of platelet transfusions) to ≥ 50,000 /µL lasting for at least 2 weeks.
Time Frame: Up to 12 weeks
Population: Participants who completed study
Measure: Number; unit: Percent of participants
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
Percent of participants | 90

8. Secondary Outcome: Median Days to Attain Complete Response
Description: The median number of days participants take to achieve a complete response as defined as a sustained improvement of platelet counts (independent of platelet transfusions) to ≥ 50,000 /µL lasting for at least 2 weeks.
Time Frame: Up to 12 weeks
Population: Participants who completed study
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
days | 30 [25 to 34]

9. Secondary Outcome: Partial Complete Response Rate
Description: The number of participants with a sustained improvement of platelet counts (independent of platelet transfusions) seen by at least a doubling of platelet count from the pretreatment thrombocytopenic level (defined as < 10000 /µL, ) or an absolute increase in platelet counts to between 30000 /µL and 50000 /µL, whichever is higher but not achieving complete response. Or if there is a need to restart eltrombopag due to drop in platelet count to below 50000 /µL following interruption of eltrombopag therapy after achieving platelet counts of > 100000 /µL on the drug.
Time Frame: Up to 12 weeks
Population: Participants who completed study
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
Participants | 0

10. Secondary Outcome: Time to Initiation of Post-remission Therapy
Description: The average number of days from the the beginning of treatment to the onset of post-remission therapy as summarized using the Kaplan-Meier method and calculated using the logrank test and proportional hazards models.
Time Frame: Up to 12 weeks
Population: as for outcome 5
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 0

11. Secondary Outcome: Rate of Refractory or Persistent Disease
Description: The number of participants with presence of morphologic evidence of disease
Time Frame: Up to 12 weeks
Population: Participants who completed study
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
Participants | 0

12. Secondary Outcome: Overall Survival (OS) - Percent of Participants Alive at Follow-up
Description: OS is defined from the day of study registration until the last follow-up or death
Time Frame: at 28 days, at 6 months and up to 5 years
Population: Participants who went on study
Measure: Number; unit: percent of participants
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
percent of participants
  28 days from start of treatment | 100
  6 months from start of treatment | 74.2

13. Secondary Outcome: Number of Participants With 3/4 Adverse Events Adverse Events, Determined According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Incidence of grade 3/4 adverse events (AE), determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
  For full list, see AE/serious adverse event (SAE) section
Time Frame: Up to 4 weeks after last dose of eltrombopag olamine
Population: Participants enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Eltrombopag Olamine)
Number analyzed (Participants) | 31
Participants
  febrile neutropenia | 1
  thromboembolic event | 1
  rash | 1
  generalized myalgias | 1
  hypokalemia & hypocalhypokalemia & hypocalcemia | 1

14. Secondary Outcome: Disease-Free Survival
Description: Calculated from the date of complete remission until relapse, the date of last follow-up, or other protocol-defined event
Time Frame: At 5 year follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events are collected for 4 weeks post intervention and mortality is monitored for up to 5 years of follow-up
Arm/Group | Supportive Care (Eltrombopag Olamine)
All-Cause Mortality (participants affected / at risk) | 8/31
Serious Adverse Events (participants affected / at risk) | 14/31
Other Adverse Events (participants affected / at risk) | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Eltrombopag Olamine) (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Cardiac troponin T increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hematuria (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Eltrombopag Olamine) (N=31)
Anemia (Blood and lymphatic system disorders) | 12 (14)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (11)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Ileus (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 4 (4)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 9 (11)
Fatigue (General disorders) | 3 (4)
Fever (General disorders) | 5 (5)
Non-cardiac chest pain (General disorders) | 2 (2)
Blood infections (Infections and infestations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 8 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (7)
Confusion (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT02071901/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT02071901/ICF_001.pdf